CLINICAL TRIAL: NCT00326586
Title: A Phase I Dose-Escalation Study of BMS-641988 in Patients With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CA185-002
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BMS 641988

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AR Antagonist (BMS-641988)

INTERVENTIONS:
Drug: AR Antagonist (BMS-641988) — Tablets, Oral, 6 Patients will be randomized in a 1:1 ratio and in a double-blinded fashion to achieve a single dose of the study drug or Placebo on C1D1. Once daily, at least 3 cycles until the disease progresses

SUMMARY:
This is a Phase I Dose-Escalation Study of BMS641988 in Patients with Castration-Resistant Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced castration-resistant prostate carcinoma with progressive disease
* At least 4 weeks must have elapsed from major surgery
* Patient must be available for follow-up
* Adequate liver and kidney function
* Adequate blood values

Exclusion Criteria:

* Uncontrolled or significant heart disease
* History of seizures
* History of head injury, loss of consciousness, or stroke
* Patients undergoing alcohol withdrawal
* Any concurrent cancer
* A serious uncontrolled medical disorder or active infection
* Inability to swallow tablets

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability and to identify a dose for Phase II evaluation | during the dose escalation phase

SECONDARY OUTCOMES:
To evaluate pharmacokinetics | throughout the study
To describe preliminary evidence of anit-tumor activity | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University Of Wisconsin Hospital And Clinics Laboratory, Madison, Wisconsin

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx